CLINICAL TRIAL: NCT05031195
Title: Preoperative Neutrophil to Lymphocyte Ratio, Platelet to Lymphocyte Ratio, and Mean Platelet Volume as Predictors of 1 Year Mortality in Patients Undergoing an Open Repair of Abdominal Aortic Aneurysms: a Retrospective Study
Brief Title: Prognostic Impact of NLR, PLR, and MPV in Patients Undergoing AAA Open Repair
Status: Completed | Type: Observational
Sponsor: Gangnam Severance Hospital (Other)
Responsible Party: Principal Investigator, Sung Yeon Ham, Associate Professor, Gangnam Severance Hospital
Other Study IDs: 3-2020-0479
Record Dates: First submitted 2021-08-29; First posted 2021-09-01 (Actual); Last update posted 2022-03-25 (Actual); Status verified 2022-03

CONDITIONS: Abdominal Aortic Aneurysm
Keywords: neutrophil to lymphocyte ratio; platelet to lymphocyte ratio; mean platelet volume; aortic surgery; abdominal aortic aneurysm.
MeSH Terms: conditions — Aortic Aneurysm, Abdominal

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- 1st tertile
  Interventions: Other: 1st tertile, 2nd tertile, 3rd tertile
- 2nd tertile
  Interventions: Other: 1st tertile, 2nd tertile, 3rd tertile
- 3rd tertile
  Interventions: Other: 1st tertile, 2nd tertile, 3rd tertile

INTERVENTIONS:
Other: 1st tertile, 2nd tertile, 3rd tertile — Patients will be divided into 3 groups according to the preoperative NLR value.

SUMMARY:
Abdominal aortic aneurysm (AAA) is a multifactorial degenerative disorder, which if untreated might lead to catastrophic complications. The treatment for AAA includes open and endovascular repair, both of which carry a significant degree of risk. Thus, researchers have performed several studies addressing simple and readily available risk stratification markers, such as complete blood count in patients undergoing open AAA repair.

The neutrophil to lymphocyte ratio (NLR) has been frequently used as a marker of systemic inflammatory response, which reflects neutrophilia and lymphopenia. The primary pathophysiology of AAA involves chronic inflammation in the aortic wall and atherosclerosis, accompanied with thrombosis. NLR was proposed as a fair indicator for poor prognosis in patients with AAA. The mean platelet volume (MPV) is the marker of platelet activation and an indicator of the activation of thrombus formation. Moreover, it is reportedly associated with the prognosis of patients with cardiovascular diseases. Moreover, the platelet to lymphocyte ratio (PLR) suggests thrombosis and inflammation and indicates a high risk of cardiovascular events in various groups of patients. The PLR is associated with poor prognosis following AAA repair. Despite accumulating evidence for the prognostic value of white blood cell counts in abdominal aortic aneurysm, few studies have investigated the value of these parameters, including NLR, MPV, and PLR, in patients undergoing AAA open repair.

The investigators aimed to investigate if preoperative neutrophil to lymphocyte ratio (NLR), platelet to lymphocyte ratio (PLR), or mean platelet volume (MPV) could be used to predict 1-year mortality in patients undergoing open abdominal aortic aneurysm (AAA) repair.

DETAILED DESCRIPTION:
The investigators will retrospectively review medical records who underwent open abdominal aortic aneurysm repair between Jan 2008 and July 2019. The investigators will divide the patients into two groups according to the occurrence of 1-yr mortality. Then the investigators compare complete blood count including NLR, PLR and MPV between the groups. Furthermore, the patient will be divided into tertiles according to the preoperative NLR, PLR, and MPV values to compare the incidence of 1-yr mortality and other morbidities. Multivariable logistic regression analysis will be performed to investigate possible prognostic factor for 1-yr mortality in these patients.

ELIGIBILITY:
Inclusion Criteria:

* patients who underwent open repair of abdominal aortic aneurysm.

Exclusion Criteria:

* patients with previous aortic repair within 6 months.
* mycotic aneurysm.
* iliac artery aneurysm.
* aorta occlusive disease.
* incomplete data.

Ages: 19 Years to 99 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients undergoing open AAA repair in university hospital.
Sampling Method: Non-Probability Sample
Enrollment: 334 (Actual)
Dates: Start 2020-01-11 (Actual); Primary Completion 2021-03-30 (Actual); Study Completion 2021-03-30 (Actual)

PRIMARY OUTCOMES:
The incidence of postoperative 1-yr mortality | 1-yr after operation
  The incidence of postoperative 1-yr mortality in patients undergoing open repair of abdominal aortic aneurysm.

CONTACTS AND LOCATIONS:
Locations (1):
- Gangnam Severance Hospital, Seoul, South Korea